CLINICAL TRIAL: NCT00079560
Title: THC and Marijuana--Effects in Individuals With HIV/AIDS
Brief Title: Comparing the Effects of Smoked and Oral Marijuana in Individuals With HIV/AIDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Jag H. Khalsa, Ph.D., National Institute on Drug Abuse, NIH
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01DA012698-01A1 (NIH)
Expanded Access: Available
Record Dates: First submitted 2004-03-09; First posted 2004-03-10 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2008-10

CONDITIONS: HIV Infections
Keywords: HIV; Marijuana; Marinol; Oral THC; Appetite; Complementary Therapies
MeSH Terms: conditions — HIV Infections; Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: dronabinol — dronabinol to prevent development of marijuana withdrawal

SUMMARY:
Smoked marijuana (MJ) and dronabinol (also known as THC or by the trade name Marinol) are used to increase appetite, food intake, and weight in patients with HIV who experience unintended weight loss. This study will compare the effects of MJ and Marinol use in marijuana smokers who are HIV infected.

DETAILED DESCRIPTION:
Little is known about the efficacy and tolerability of oral THC versus smoked MJ in a clinically relevant population. Additionally, it is not clear how THC's effects vary as a function of the duration of treatment or the patient's current patterns of smoked MJ use. This study directly compares 3 doses of smoked marijuana and 3 doses of Marinol across a range of behavioral measures in HIV infected marijuana smokers.

Outcome measures will include analysis of food intake, body composition, mood, physical symptoms (e.g., nausea, stomach pain), psychomotor task performance, and sleep.

ELIGIBILITY:
Inclusion Criteria

* HIV infected
* Smoke marijuana
* Taking HIV medications

Exclusion criteria

* Naive marijuana smokers
* People with history of respiratory/pulmonary disease

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2001-12; Primary Completion 2004-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
daily caloric intake | daily measure of colories

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States